CLINICAL TRIAL: NCT01581229
Title: Early Use of Noninvasive Positive Pressure Ventilation for Intro-pulmonary Acute Lung Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Chen Wang, vice president, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012BAI05B00
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Acute Lung Injury
Keywords: ALI;noninvasive positive pressure ventilation
MeSH Terms: conditions — Acute Lung Injury | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPPV (Experimental)
  Interventions: Procedure: noninvasive positive pressure ventilation
- Control (Active Comparator)
  Interventions: Procedure: oxygen therapy

INTERVENTIONS:
Procedure: noninvasive positive pressure ventilation — Patients in the NPPV group are ventilated using the CPAP or bilevel positive airways pressure S/T mode.
  Arms: NPPV
Procedure: oxygen therapy — In the control group, Venturi masks are used to maintain SpO2 at 92% to 96% by adjusting the oxygen flow rates.
  Arms: Control

SUMMARY:
To assess the safety and efficacy of noninvasive positive pressure ventilation for patients with intro-pulmonary pulmonary acute lung injury and compare this with high-concentration oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

1. acute onset;
2. a clinical presentation of respiratory distress;
3. arterial oxygen tension/inspired oxygen fraction (PaO2/FIO2) < 300 mmHg but > 200 mmHg while breathing oxygen delivered by a conventional Venturi device at a maximum concentration (50%);
4. presence of bilateral pulmonary infiltrates on posteroanterior chest radiograph;
5. no evidence of left heart failure as assessed by echocardiography and/or a pulmonary artery wedge pressure of <18 mm Hg.
6. the cause of ALI is consider to be intro-pulmonary.

Exclusion Criteria:

1. age <18 yrs;
2. Glasgow Coma Scale < 11;
3. airway or facial injury;
4. pneumothorax or pneumomediastinum;
5. unable to spontaneously clear secretions from the airways;
6. cardiogenic shock or severe hemodynamic instability (systolic blood pressure <90 mmHg associated with decreased urinary output (<20 mL.h-1) despite fluid repletion and use of vasoactive agents) of other causes;
7. severe ventricular arrhythmia or unstable myocardial ischemia;
8. severe organ dysfunction (Sequential Organ Failure Assessment score > 3);
9. end-stage patients who were expected to survive < 6 months;
10. severe abdominal distension;
11. refusal to receive NPPV;
12. the cause of ALI is consider to be extrapulmonary;
13. unable to cooperate with NPPV application;
14. active upper gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
numbers of patients who met the intubation criteria | 1 year
the numbers of patients who are actually intubated | 1 year

SECONDARY OUTCOMES:
inhospital mortalities | 1 year
intensive care unit mortalities | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, MD, PHD, Principal Investigator — Beijing Hospital of the Ministry of Health; Beijing Institute of Respiratory Medicine
Locations (1):
- Beijing Hospital of the Ministry of Health, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] He H, Sun B, Liang L, Li Y, Wang H, Wei L, Li G, Guo S, Duan J, Li Y, Zhou Y, Chen Y, Li H, Yang J, Xu X, Song L, Chen J, Bao Y, Chen F, Wang P, Ji L, Zhang Y, Ding Y, Chen L, Wang Y, Yang L, Yang T, Weng H, Li H, Wang D, Tong J, Sun Y, Li R, Jin F, Li C, He B, Sun L, Wang C, Hu M, Yang X, Luo Q, Zhang J, Tan H, Wang C; ENIVA Study Group. A multicenter RCT of noninvasive ventilation in pneumonia-induced early mild acute respiratory distress syndrome. Crit Care. 2019 Sep 4;23(1):300. doi: 10.1186/s13054-019-2575-6. PMID 31484582